CLINICAL TRIAL: NCT05439226
Title: Liver Fat as a Dietary Target of the Chinese Medical Nutrition Therapy (CMNT) Diet for Treating Type 2 Diabetes With Nonalcoholic Fatty Liver Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State Key Laboratory of Subhealth Intervention Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Version 2.0
Record Dates: First submitted 2022-06-21; First posted 2022-06-30 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes with NAFLD; CMNT diet
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CMNT diet (Experimental): The CMNT group was instructed to consumed the provided CMNT diet consisting of 6 cycles of 5 consecutive days followed by 10 days of ad libitum food consumption. Participants received a 917 kcal/day preprepared human CMNT diet (44.75% carbohydrate, 9.1% protein and 46.15% fat) for 5 consecutive days per cycle
  Interventions: Other: CMNT diet
- Usual Care (No Intervention): Dietary recommendations based on the Guideline for the prevention and treatment of type 2 diabetes mellitus in China (2020 edition) as the control group

INTERVENTIONS:
Other: CMNT diet — Hypocaloric CMNT diet plan: A diet plan with intermittent use of enriched traditional-Chinese-medicinal-foods CMNT diet
  Arms: CMNT diet

SUMMARY:
Type 2 diabetes (T2D) represents a serious public health problem. Patients with T2D and non-alcoholic fatty liver disease(NAFLD) demonstrate a poor metabolic profile and increase mortality compared with patients with only NAFLD or T2D. Nutritional intervention is the most basic treatment for T2D. Previous study showed that a Chinese medical nutrition therapy (CMNT) diet, which intermittent use of low-calorie medicinal food, has a glucose-lowering effect in T2D. This study aims to investigate the effect of a Chinese medical nutrition therapy (CMNT) diet accompanied by intermittent energy restriction on reducing liver fat and glycated hemoglobin (HbA1c) in patients with T2D and NAFLD.

DETAILED DESCRIPTION:
Diet composition of CMNT is a multicomponent Chinese medicinal food, which mainly enriched with whole grains and edible medicine and food homologous (MFH) plants such as Rhizoma Dioscoreae, Momordica Grosvenori, Folium Mori, Radix Puerariae, Fructus lycii, Poria cocos that meets the requirements of a food for special medical purpose. The CMNT group was instructed to consumed the provided CMNT diet consisting of 6 cycles of 5 consecutive days followed by 10 days of ad libitum food consumption. Participants received a 917 kcal/day preprepared human CMNT diet (44.75% carbohydrate, 9.1% protein and 46.15% fat) for 5 consecutive days per cycle. CMNT diet is composed of four ready-to-consume prepared foods including composite nutritional rice, solids beverages, meal replacement biscuit and fruit and vegetable gruel mainly from wholegrains and traditional Chinese medicinal food plants. The intervention lasted for 3 months (6 cycles) and follow-up measurements will be performed in all subjects after 3-months from end of the intervention. The glucose-lowering medication use of participants strictly implemented by their physician according to the diabetes medications management protocol. Treatment-as-usual control group continued to be given standard medication and dietary advice by their physician followed guidelines for the prevention and control of T2D in China.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with type 2 diabetes and NAFLD
* Age between 18 and 75 years
* BMI between 18.0 and 35.0 kg/m2
* Weight stable for at least 3 months prior to the study (gain or loss < 4 kg)
* Stable treatment for at least 3 months with 1-3 oral antidiabetic medications (with or without insulin therapy), or not yet received antidiabetic medication prior to the beginning of the study
* Able to give written informed consent

Exclusion Criteria:

* Self-reported a food allergy
* Alcohol abuse in the last 3 months (alcohol intake greater than 20 g per day for women; Alcohol intake for men greater than 40 g per day)
* Other liver diseases such as chronic hepatitis B and C, autoimmune hepatitis, primary biliary cirrhosis, hemochromatosis, nodular regenerative hyperplasia and focal nodular hyperplasia
* Scheduled to be hospitalized for any surgical treatment during screening
* Pregnant or planning of pregnancy during the study
* Inability, physically or mentally, to adhere the procedures required by the study protocol
* Level 3 hypoglycemic events (at least 3 times) occurring within the 90 days prior to screening
* Hospitalization or emergency department visit for hyperglycemia, diabetic ketoacidosis, lactic acidosis, hyperosmolar nonketotic coma, or diabetes
* History of cancer within the past 5 years
* Acute coronary or cerebrovascular event in the past 90 days, or heart failure
* Hemorrhagic or ischemic stroke within the last 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2026-05-05 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
Controlled attenuation parameter (CAP) value by transient elastography | 3, 6, 12, 24 months
  The CAP score, which be measured by FibroScan, will be used to quantify and detect liver fat. CAP < 238 dB/m indicated no hepatic steatosis, 238 ≤ CAP ≤ 259 dB/m denoted mild steatosis, 260 ≤ CAP ≤291 dB/m indicated moderate steatosis, and CAP > 291 dB/m denoted severe steatosis.
HbA1C | 3, 6, 12, 24 months
  Blood test to measure glucose control

SECONDARY OUTCOMES:
Fatty liver index (FLI) | 3, 6, 12, 24 months
  FLI will also be applied to quantify the degree of steatosis of patients with type 2 diabetes and NAFLD. FLI values < 30 rule out liver steatosis, whereas FLI ≥ 60 confirmed NAFLD with a specificity of 61%.
Hepatic steatosis index (HSI) | 3, 6, 12, 24 months
  HSI will also be applied to quantify the degree of steatosis of patients with type 2 diabetes and NAFLD. HSI values < 30 excludes NAFLD with a sensitivity of 93.1%, while values > 36 detected NAFLD with a specificity of 92.4%.
Liver stiffness measurement (LSM) value by transient elastography | 3, 6, 12, 24 months
  Liver fibrosis will be assessed by using a non-invasive vibration-controlled transient elastography to estimate LSM. A median LSM ≥ 8.2 kPa was considered indicative of significant fibrosis (≥ F2), whereas LSM ≥ 9.7 kPa was considered indicative of advanced (≥ F3) fibrosis, whereas LSM ≥ 13.6 kPa was considered indicative of cirrhosis (F4).
Fibrosis-4 index (FIB-4) | 3, 6, 12, 24 months
  The FIB-4 index, a non-invasive measurement, will be used to evaluate the degree of liver fibrosis. The FIB-4 index <1.45 had a negative predictive value of 94.7% to exclude progressive fibrosis, whereas FIB-4 index >3.25 was considered advanced fibrosis or cirrhosis.
NAFLD fibrosis score (NFS) | 3, 6, 12, 24 months
  Degree of liver fibrosis will also be assessed by NFS.The probability of advanced liver fibrosis was classified into three groups: high NFS (NFS > 0.676), intermediate NFS (NFS: -1.455 to 0.676, or 0.120 to 0.676 if age > 65), or low NFS (NFS < -1.455, or < 0.120 if age > 65) .
Liver function test | 3, 6, 12, 24 months
  γ-glutamyl transferase (γ-GGT), alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP) and ect will be assessed.
Blood glucose | 3, 6, 12, 24 months
  Fasting plasma glucose (FPG) and postprandial 2-hour plasma glucose (2 h-PG)
Blood lipid | 3, 6, 12, 24 months
  triglyceride, total cholesterol, low-density lipoprotein cholesterol (LDL-C) and high-density lipoprotein-cholesterol (HDL-C)
Insulin | 3, 6, 12, 24 months
  Glucose homeostasis
HOMA-IR | 3, 6, 12, 24 months
  Fasting glucose times fasting insulin divided by 22.5
IGF-1 | 3, 6, 12, 24 months
  Glucose homeostasis
Body mass index | 3, 6, 12, 24 months
  Body mass in kilograms divided by height in meters squared.
waist-to-hip ratio | 3, 6, 12, 24 months
  Waist circumference in centimeter divided by height in centimeter.
Blood pressure | 3, 6, 12, 24 months
  Systolic blood pressure and diastolic blood pressure.
Energy intake | 3, 6, 12, 24 months
  3-day diet record and Food Frequency Questionnaire
Macronutrient intake | 3, 6, 12, 24 months
  3-day diet record and Food Frequency Questionnaire
Sleep quality | 3, 6, 12, 24 months
  Pittsburgh Sleep Quality Index Questionnaire
Physical activity | 3, 6, 12, 24 months
  International Physical Activity Questionnaire
Self-reported depressive symptoms | 3, 6, 12, 24 months
  Patient Health Questionnaire 9
Anxiety symptoms | 3, 6, 12, 24 months
  Generalized Anxiety Disorder scale
Social support | 3, 6, 12, 24 months
  Social Support Rate Scale
Reduction in glucose-lowering medication | 3, 6, 12, 24 months
  Reduction in total dose of glucose-lowering medications
Fecal microbiota profile | 3, 6, 12, 24 months
  Fecal samples will be collected and will be sequenced.
Metabolomics | 3, 6, 12, 24 months
  Blood, fecal and urine samples will be collected and metabolites will be analyzed through a metabolomics approach.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Physical Examination Center of Gezhouba central hospital of Sinopharm, Yichang, Hubei
  - Hunan Shanshui physical examination center, Changsha, Hunan
  - Jinheyuan Outpatient Department, National Sub-health Intervention Technology Achievement Application Center, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Luo W, Xiao Z, Yang X, Wu R, Li J, Yu Z, Guo S, Nie B, Liu D. Liver fat as a dietary target by Chinese Medical Nutrition Therapy (CMNT) diet for treating type 2 diabetes with non-alcoholic fatty liver disease: study protocol for a randomised controlled trial. BMJ Open. 2024 Apr 29;14(4):e081263. doi: 10.1136/bmjopen-2023-081263. PMID 38684277

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-12): https://cdn.clinicaltrials.gov/large-docs/26/NCT05439226/Prot_SAP_000.pdf